CLINICAL TRIAL: NCT03737240
Title: A Randomized Controlled Trial Comparing the Safety and Efficacy of IDegLira Versus Basal Bolus in Patients With Poorly Controlled Type 2 Diabetes
Brief Title: IDegLira HIGH Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Rodolfo Galindo, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00104726
Record Dates: First submitted 2018-11-08; First posted 2018-11-09 (Actual); Results first posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Diabetes Mellitus
Keywords: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — IDegLira; insulin degludec; Liraglutide; Insulin Aspart

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1 to 1 ratio to receive the study treatment or standard of care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IDegLira (Experimental): Participants in this group will receive IDegLira (with metformin, unless contraindicated) for 26 weeks.
  Interventions: Drug: IDegLira
- Basal-Bolus Insulin (Active Comparator): Participants in this group will receive basal-bolus insulin (with metformin, unless contraindicated) for 26 weeks. The basal-bolus insulin regimen includes Insulin Degludec (U-100) and Insulin Aspart.
  Interventions: Drug: Insulin Degludec (U-100); Drug: Insulin Aspart

INTERVENTIONS:
Drug: IDegLira — Participants in this study arm will discontinue all other diabetes medications, except for metformin which will be continued at prescribed dose (unless contraindicated). IDegLira will be given once daily, at the same time of the day with or without food for 26 weeks. IDegLira will be titrated until the maximum dose is reached, up to the target fasting blood glucose of 70 to 100 milligrams per deciliter (mg/dL).
  Other Names: Xultophy 100/3.6; insulin degludec; liraglutide
  Arms: IDegLira
Drug: Insulin Degludec (U-100) — Participants in the basal-bolus insulin study arm will discontinue all other diabetes medications, except for metformin which will be continued at the prescribed dose (unless contraindicated). Insulin Degludec (U-100) will be given once daily at the same time for 26 weeks. The dose will be titrated up to the fasting blood glucose target of 70 to 100 mg/dL, with no maximum dose.
  Other Names: Tresiba FlexTouch
  Arms: Basal-Bolus Insulin
Drug: Insulin Aspart — Participants in the basal-bolus insulin study arm will discontinue all other diabetes medications, except for metformin which will be continued at the prescribed dose (unless contraindicated). Insulin aspart will be taken before meals with a titration schedule and dose adjustment protocol to target pre-meal blood glucose level of 70 to 100 mg/dL.
  Other Names: NovoLog
  Arms: Basal-Bolus Insulin

SUMMARY:
Basal-bolus insulin therapy is recommended for patients with poorly controlled type 2 diabetes (T2D) and HbA1c >9%. However, basal-bolus insulin is labor intensive and associated with increased risk of hypoglycemia, glycemic variability, weight gain and poor compliance. Thus, there is a critical need for a simpler treatment regimen that could overcome these limitations. IDegLira, a fixed-ratio combination (FRC) therapy consisting of insulin degludec and liraglutide, is an attractive option for this population given its proven benefits on glycemic control, weight and compliance. This study aims to show that a simpler regimen using a novel FRC agent (IDegLira) can improve glycemic control, decrease hypoglycemia, reduce the burden of diabetes care, and improve satisfaction/adherence in patients with poorly controlled T2D with HbA1c between ≥ 9-12%. This open-label, treat-to- target, two-arm parallel, controlled trial will randomize participants with T2D and HbA1c ≥ 9%, treated with oral anti-diabetic agents and/or basal insulin therapy to lDegLira or basal-bolus insulin for 26 weeks.

DETAILED DESCRIPTION:
Extensive literature has shown that persistent hyperglycemia is associated with short- and long-term complications. Sustained hyperglycemia, also known as glucotoxicity, leads to progressive loss of beta-cell function and is considered a key pathophysiological process in the development of type 2 diabetes (T2D). Patients with severe hyperglycemia may respond poorly to oral anti-diabetic agents (OAD) alone initially and frequently require insulin to achieve glycemic targets. Current guidelines recommend to initiate therapy with basal insulin and progressively step up to basal-bolus insulin in patients with high HbA1c >9%, particularly if symptomatic or with catabolic symptoms.

A basal-bolus insulin regimen increases the risk of hypoglycemia, weight gain and glycemic variability, which are limiting factors in achieving glycemic targets. A basal-bolus insulin regimen is also labor intensive and often requires multiple daily injections, further increasing the burden of diabetes care and decreasing patient adherence. In contrast, simplified treatment plans may improve adherence, leading to glycemic targets achievement. Thus, there is a critical need for simpler regimens that could overcome clinical inertia, improve patient adherence, and decrease glycemic variability in patients with poorly controlled type 2 diabetes. This prospective randomized control trial will compare IDegLira to basal-bolus insulin regimen in achieving glycemic control, while reducing hypoglycemia, glycemic variability, and weight gain in patients with uncontrolled T2D and HbA1c ≥9%.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes, diagnosed for ≥ 6 months
* HBA1c ≥ 9% - 15%
* Previously treated with oral antidiabetic agents, including metformin, sulfonylurea, repaglinide/nateglinide, pioglitazone, dipeptidyl peptidase-4 (DPP4), inhibitors, SGLT2 inhibitors, (monotherapy + basal insulin) or in combination therapy (2-3 agents), and/or on basal insulin (neutral protamine hagedorn (NPH), detemir or glargine U100) at a total daily dose (TDD) 20-50 units (stable doses of metformin and basal insulin for at least 90 days, defined as up to ±10% variability)
* Body mass index (BMI) ≤ 45 Kg/m2

Exclusion Criteria:

* Subjects with type 1 diabetes or latent autoimmune diabetes of adults (LADA) (positive glutamic acid decarboxylase (GAD-65) antibody and/or ketones)
* Subjects with a BG > 400 mg/dL during the screening visit and laboratory evidence of diabetic ketoacidosis
* Previous treatment with glucagon-like peptide-1 (GLP-1) agonists (during prior 3 months)
* Previous treatment with basal-bolus insulin (within prior 3 months)
* Recurrent severe hypoglycemia or known hypoglycemia unawareness.
* Personal or family history of medullary thyroid cancer or multiple endocrine neoplasia 2
* Patients with acute or chronic pancreatitis, pancreatic cancer
* Patients with clinically significant hepatic disease (cirrhosis, jaundice, end-stage liver disease) or significantly impaired renal function (GFR < 30 ml/min).
* Treatment with oral or injectable corticosteroid (equivalent or higher than prednisone 5 mg/day), parenteral nutrition and immunosuppressive treatment.
* Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study
* Hypersensitivity to study drugs
* Participating in another investigational drug trial
* The receipt of any investigational drug (within 3 months) prior to this trial.
* Previously randomized in this trial
* Heart Failure New York Heart Association (NYHA) class 4 or uncontrolled hypertension (blood pressure > 180/110 mmHg)
* Female subjects who are pregnant or breast-feeding at time of enrollment into the study
* Females of childbearing potential who are not using adequate contraceptive methods (as required by local law or practice)
* Known or suspected allergy to trial medications (degludec, liraglutide, aspart), excipients, or related products.
* Subjects could be excluded based on PI's discretion
* Unable to comply with trial protocol, and/or at investigator discretion
* Patients receiving treatment for active diabetic retinopathy or with proliferative retinopathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Galindo, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Grady Health System, Atlanta, Georgia
  - Emory Clinic, Atlanta, Georgia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IDegLira | Basal-Bolus Insulin
Started | 72 | 73
Completed | 56 | 58
Not Completed | 16 | 15
Not completed — Lost to Follow-up | 16 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDegLira | Basal-Bolus Insulin | Total
Number analyzed (Participants) | 72 | 73 | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (10.1) | 53.8 (9.7) | 54.21 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 35 | 63
  Male | 44 | 38 | 82
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 63 | 61 | 124
  White | 3 | 7 | 10
  More than one race | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 72 | 73 | 145

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin A1c (HbA1c)
Description: HbA1c will be compared between study groups. HbA1c measures the average percentage of blood sugar over the past 2 to 3 months and HbA1c can reduce with management of diabetes through diet, exercise, and medication. HbA1c levels below 5.7% are considered normal. Persons with values between 5.7% and 6.4% are considered at high risk of developing diabetes while those with values of 6.5% and above are diagnosed with diabetes. Persons with diabetes aim to get their HbA1c in the range of 7.0 to 7.5% or lower, with below 7.0% being preferable.
Time Frame: Baseline, Week 26
Population: Number of patients analyzed include participants that completed the visit and had a valid HbA1c result.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | IDegLira | Basal-Bolus Insulin
Number analyzed (Participants) | 56 | 58
percentage of HbA1c | -3.18 (2.29) | -3.00 (1.79)

2. Secondary Outcome: Average Fasting Blood Glucose
Description: Mean fasting blood glucose will be compared between study arms. Participants will perform an 8-point, self-monitored blood glucose (SMBG) check by testing their blood sugar at 8 different time points. The measurement taken before breakfast is used to assess fasting blood glucose. For people without diabetes, fasting blood glucose is typically between 70-100 mg/dL while fasting blood glucose for those with diabetes is in the range of 70-130 mg/dL.
Time Frame: Week1, Week 12, Week 26
Population: Number of participants analyzed include total patients that completed each study visit and provided data for each study visit.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | IDegLira | Basal-Bolus Insulin
Number analyzed (Participants) | 72 | 73
mg/dL
  Baseline (Week 1) | 202.37 (63.73) | 206.53 (58.04)
  Week 12: number analyzed (Participants) | 61 | 63
  Week 12 | 131.94 (45.59) | 125.18 (29.29)
  Week 26: number analyzed (Participants) | 56 | 58
  Week 26 | 143.31 (89.55) | 143.14 (62.81)

3. Secondary Outcome: Average Daily Blood Glucose
Description: Mean daily blood glucose will be compared between study arms. Participants will perform an 8-point, self-monitored blood glucose (SMBG) check by testing their blood sugar at 8 different time points. Blood glucose levels vary depending on when and what food has been consumed. A blood glucose level taken regardless of timing of meals of greater than 200 mg/dL often indicates diabetes. Blood glucose decreases with improved diabetes management.
Time Frame: Week1, Week 12, Week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | IDegLira | Basal-Bolus Insulin
Number analyzed (Participants) | 72 | 73
mg/dL
  Week 1 (Baseline) | 220.81 (64.43) | 225.18 (65.74)
  Week 12: number analyzed (Participants) | 61 | 63
  Week 12 | 143.80 (47.72) | 135.08 (33.51)
  Week 26: number analyzed (Participants) | 56 | 58
  Week 26 | 134.59 (36.35) | 144.25 (40.70)

4. Secondary Outcome: Participants With HbA1c <7.0% and no Hypoglycemia
Description: Percent of study participants experiencing HbA1c <7.0% and no hypoglycemia will be compared between groups. Persons with diabetes aim to get their HbA1c in the range of 7.0 to 7.5% or lower, with below 7.0% being preferable. Hypoglycemia is defined as a blood glucose level of < 70 mg/dL.
Time Frame: Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | IDegLira | Basal-Bolus Insulin
Number analyzed (Participants) | 72 | 73
Participants | 19 | 6

5. Secondary Outcome: Participants With HbA1c <7.0% and no Weight Gain and no Hypoglycemia
Description: Percent of study participants reaching A1c < 7% without weight gain and no hypoglycemia will be compared between groups. Weight control is typically important in persons with type 2 diabetes and basal-bolus insulin is associated with weight gain. Persons with diabetes aim to get their HbA1c in the range of 7.0 to 7.5% or lower, with below 7.0% being preferable. Hypoglycemia is defined as a blood glucose level of < 70 mg/dL.
Time Frame: Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | IDegLira | Basal-Bolus Insulin
Number analyzed (Participants) | 72 | 73
Participants | 8 | 1

6. Secondary Outcome: Participants With HbA1c <7.5% and no Weight Gain and no Hypoglycemia
Description: Percent of study participants reaching A1c < 7.5% without weight gain and no hypoglycemia will be compared between groups. Weight control is typically important in persons with type 2 diabetes and basal-bolus insulin is associated with weight gain. Persons with diabetes aim to get their HbA1c in the range of 7.0 to 7.5% or lower, with below 7.0% being preferable. Hypoglycemia is defined as a blood glucose level of < 70 mg/dL.
Time Frame: Week 26
Population: This outcome include participants with a baseline HbA1c <7.5%.
Measure: Number; unit: percentage of participants
Arm/Group | IDegLira | Basal-Bolus Insulin
Number analyzed (Participants) | 56 | 57
percentage of participants | 19.6 | 5.2

7. Secondary Outcome: Participants With HbA1c >10% Achieving HbA1c <7.5%
Description: Percent of study participants with baseline HbA1c >10% reaching A1c < 7.5% will be compared between study groups. HbA1c measures the average percentage of blood sugar over the past 2 to 3 months and HbA1c can reduce with management of diabetes through diet, exercise, and medication. HbA1c levels below 5.7% are considered normal. Persons with values between 5.7% and 6.4% are considered at high risk of developing diabetes while those with values of 6.5% and above are diagnosed with diabetes. Persons with diabetes aim to get their HbA1c in the range of 7.0 to 7.5% or lower, with below 7.0% being preferable.
Time Frame: Baseline, Week 26
Population: This outcome includes participants with a baseline HbA1c >10%.
Measure: Number; unit: percentage of participants
Arm/Group | IDegLira | Basal-Bolus Insulin
Number analyzed (Participants) | 44 | 48
percentage of participants | 56.8 | 37.5

8. Secondary Outcome: Participants With HbA1c >10% Achieving HbA1c <8.0%
Description: Percent of study participants with baseline HbA1c >10% reaching A1c < 8.0% will be compared between study groups. HbA1c measures the average percentage of blood sugar over the past 2 to 3 months and HbA1c can reduce with management of diabetes through diet, exercise, and medication. HbA1c levels below 5.7% are considered normal. Persons with values between 5.7% and 6.4% are considered at high risk of developing diabetes while those with values of 6.5% and above are diagnosed with diabetes. Persons with diabetes aim to get their HbA1c in the range of 7.0 to 7.5% or lower, with below 7.0% being preferable.
Time Frame: Baseline, Week 26
Population: This outcome includes study participants with baseline HbA1c >10%.
Measure: Number; unit: percentage of participants
Arm/Group | IDegLira | Basal-Bolus Insulin
Number analyzed (Participants) | 44 | 48
percentage of participants | 61.4 | 45.8

9. Secondary Outcome: Participants With HbA1c >11% Achieving HbA1c <7.5%
Description: Percent of study participants with baseline HbA1c >11% reaching A1c < 7.5% will be compared between study groups. HbA1c measures the average percentage of blood sugar over the past 2 to 3 months and HbA1c can reduce with management of diabetes through diet, exercise, and medication. HbA1c levels below 5.7% are considered normal. Persons with values between 5.7% and 6.4% are considered at high risk of developing diabetes while those with values of 6.5% and above are diagnosed with diabetes. Persons with diabetes aim to get their HbA1c in the range of 7.0 to 7.5% or lower, with below 7.0% being preferable.
Time Frame: Baseline, Week 26
Population: This outcome includes study participants with baseline HbA1c >11%.
Measure: Number; unit: percentage of participants
Arm/Group | IDegLira | Basal-Bolus Insulin
Number analyzed (Participants) | 25 | 27
percentage of participants | 52.0 | 25.9

10. Secondary Outcome: Participants With HbA1c >11% Achieving HbA1c <8.0%
Description: Percent of study participants with baseline HbA1c >11% reaching A1c < 8.0% will be compared between study groups. HbA1c measures the average percentage of blood sugar over the past 2 to 3 months and HbA1c can reduce with management of diabetes through diet, exercise, and medication. HbA1c levels below 5.7% are considered normal. Persons with values between 5.7% and 6.4% are considered at high risk of developing diabetes while those with values of 6.5% and above are diagnosed with diabetes. Persons with diabetes aim to get their HbA1c in the range of 7.0 to 7.5% or lower, with below 7.0% being preferable.
Time Frame: Baseline, Week 26
Population: This outcome includes study participants with baseline HbA1c >11%.
Measure: Number; unit: percentage of participants
Arm/Group | IDegLira | Basal-Bolus Insulin
Number analyzed (Participants) | 25 | 27
percentage of participants | 60.0 | 29.6

11. Secondary Outcome: Participants With HbA1c <7.0% and no Weight Gain
Description: Percent of study participants reaching A1c < 7% without weight gain will be compared between groups.
Time Frame: Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | IDegLira | Basal-Bolus Insulin
Number analyzed (Participants) | 72 | 73
Participants | 13 | 3

12. Secondary Outcome: Participants With HbA1c <7.0% and no Hypoglycemia
Description: Percent of study participants reaching A1c < 7% without hypoglycemia will be compared between groups. Hypoglycemia is defined as a blood glucose level of < 70 mg/dL.
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | IDegLira | Basal-Bolus Insulin
Number analyzed (Participants) | 72 | 73
Participants | 21 | 8

13. Secondary Outcome: Number of Participants With Documented Symptomatic Hypoglycemic Events
Description: Documented symptomatic hypoglycemia is defined as an event with typical symptoms of hypoglycemia accompanied by SMBG <70 mg/dL or continuous glucose monitoring (CGM) < 54 mg/dL that occurs at any time of the day. Number of participants with documented hypoglycemic events will be compared between study groups.
Time Frame: Baseline through Week 26
Population: CGM hypoglycemia BG < 54 mg/dL was reported only in participants who did not have any issues with the CGM device.
Measure: Number; unit: participants
Arm/Group | IDegLira | Basal-Bolus Insulin
Number analyzed (Participants) | 72 | 73
participants
  Hypoglycemia < 70 mg/dL | 20 | 35
  Hypoglycemia < 54 mg/dL by CGM: number analyzed (Participants) | 40 | 37
  Hypoglycemia < 54 mg/dL by CGM | 21 | 26

14. Secondary Outcome: Asymptomatic Hypoglycemic Events
Description: Asymptomatic hypoglycemia is defined as no typical symptoms reported by the study participant but detected by SMBG <70 mg/dL or continuous glucose monitoring (CGM) < 54 mg/dL. Incidence of asymptomatic hypoglycemic events will be compared between study groups.
Time Frame: Baseline through Week 26
Population: Data for this outcome was not collected. Participants did not record details about symptoms when providing the blood glucose records.
Arm/Group | IDegLira | Basal-Bolus Insulin
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Number of Participants With Severe Hypoglycemic Events
Description: Severe hypoglycemia is defined as severe cognitive impairment requiring assistance from another person. Number of participants with severe hypoglycemic events will be compared between study groups.
Time Frame: Baseline through Week 26
Population: Participants who reported any BG<54 mg/dL during study participation up to 6 months
Measure: Number; unit: participants
Arm/Group | IDegLira | Basal-Bolus Insulin
Number analyzed (Participants) | 72 | 73
participants | 7 | 14

16. Secondary Outcome: Nocturnal Symptomatic Hypoglycemic Events
Description: Nocturnal symptomatic hypoglycemia is defined as an event with typical symptoms of hypoglycemia accompanied by SMBG <70 mg/dL or continuous glucose monitoring (CGM) < 54 mg/dL that occurs between midnight and 5:59 am. Incidence of nocturnal symptomatic hypoglycemic events will be compared between study groups.
Time Frame: Baseline through Week 26
Measure: Mean (Standard Deviation); unit: Number of events
Arm/Group | IDegLira | Basal-Bolus Insulin
Number analyzed (Participants) | 72 | 73
Number of events | 0.15 (1.30) | 0.16 (0.65)

17. Secondary Outcome: Nocturnal Asymptomatic Hypoglycemic Events
Description: Nocturnal asymptomatic hypoglycemia is defined as SMBG <70 mg/dL or continuous glucose monitoring (CGM) < 54 mg/dL between midnight and 5:59 am. Incidence of nocturnal asymptomatic hypoglycemic events will be compared between study groups.
Time Frame: Baseline through Week 26
Measure: Mean (Standard Deviation); unit: Number of events
Arm/Group | IDegLira | Basal-Bolus Insulin
Number analyzed (Participants) | 72 | 73
Number of events | 4.81 (7.85) | 3.45 (6.30)

18. Secondary Outcome: Percentage of Time With Interstitial Glucose <70 mg/dL
Description: Percentage of time with a interstitial glucose level below 70 mg/dL as obtained by CGM will be compared between study groups.
Time Frame: Baseline through Week 26
Population: Number of participants analyzed include total patients that completed the study visit and provided CGM data.
Measure: Mean (Standard Deviation); unit: % of time
Arm/Group | IDegLira | Basal-Bolus Insulin
Number analyzed (Participants) | 36 | 43
% of time | 2.67 (7.08) | 1.23 (2.82)

19. Secondary Outcome: Percentage of Time With Interstitial Glucose <54 mg/dL
Description: Percentage of time with a interstitial glucose level below <54 mg/dL as obtained by CGM will be compared between study groups.
Time Frame: Baseline through Week 26
Population: Number of participants analyzed include total patients that completed the study visit and provided CGM data.
Measure: Mean (Standard Deviation); unit: % of time
Arm/Group | IDegLira | Basal-Bolus Insulin
Number analyzed (Participants) | 36 | 43
% of time | 0.31 (1.22) | 0.72 (2.48)

20. Secondary Outcome: Percentage of Time With Interstitial Glucose Between 70 and 180 mg/dL
Description: Percentage of time with interstitial glucose in the range of 70-180 mg/dL as measured by CGM will be compared between study groups.
Time Frame: Baseline through Week 26
Population: Number of participants analyzed include total patients that completed the study visit and provided CGM data.
Measure: Mean (Standard Deviation); unit: % of time
Arm/Group | IDegLira | Basal-Bolus Insulin
Number analyzed (Participants) | 36 | 43
% of time | 38.39 (30.69) | 31.17 (29.00)

21. Secondary Outcome: Glycemic Variability
Description: Glycemic variability will be assessed with continuous glucose monitoring (CGM). It will be calculated using CGM and Standard Deviation.
Time Frame: Week1, Week 12, Week 26
Population: This analyses included participants that had valid CGM data at each study visit.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | IDegLira | Basal-Bolus Insulin
Number analyzed (Participants) | 51 | 61
mg/dl
  CGM Week 1 | 50.5 (14.6) | 51.6 (13.4)
  CGM Week 12: number analyzed (Participants) | 40 | 37
  CGM Week 12 | 41.8 (14.8) | 47.1 (15.4)
  CGM Week 26: number analyzed (Participants) | 36 | 43
  CGM Week 26 | 43.6 (14.8) | 48.4 (16.2)

22. Secondary Outcome: Diabetes Treatment Satisfaction Questionnaire - Status (DTSQs) Score
Description: Treatment satisfaction will be assessed with the DTSQs. The DTSQs contains eight items scored on a seven-point scale where 0 = very dissatisfied and 6 = very satisfied. The satisfaction score is obtained by summing responses to yield a total score between 0 to 48. Higher scores indicate higher satisfaction with diabetes treatment.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDegLira | Basal-Bolus Insulin
Number analyzed (Participants) | 72 | 73
score on a scale
  Baseline | 26.00 (8.06) | 29.07 (6.76)
  Follow up at 24 weeks | 33.15 (3.93) | 33.94 (2.58)

23. Secondary Outcome: Diabetes Treatment Satisfaction Questionnaire - Change (DTSQc) Score
Description: Satisfaction with the study treatment will be assessed with items 1, 4, 5, 6, 7, and 8 the DTSQc. Items are rated on a scale of -3 (much less satisfied compared to prior treatment) to 3 (much more satisfied compared to prior treatment). Total scores for these three items range from -18 to +18 with higher scores indicating greater satisfaction with the study treatment compared to their prior treatment.
Time Frame: Week 26
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDegLira | Basal-Bolus Insulin
Number analyzed (Participants) | 72 | 73
score on a scale | 15.55 (4.68) | 15.77 (3.13)

24. Secondary Outcome: Treatment-Related Impact Measures for Diabetes (TRIM-D) Survey Score
Description: Satisfaction with the study treatment will be assessed with the TRIM-D survey. TRIM-D includes 28 items that are scored on a scale from 1 to 5. Total scores are transformed to a scale of 0 to 100 where higher scores indicate increased satisfaction.
Time Frame: Baseline, Week 12, Week 26
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDegLira | Basal-Bolus Insulin
Number analyzed (Participants) | 72 | 73
score on a scale
  Baseline | 14.94 (2.29) | 15.37 (2.61)
  3 months follow up | 14.82 (1.70) | 15.29 (2.46)
  6 months follow up | 15.19 (1.88) | 15.29 (1.88)

25. Secondary Outcome: Number of Emergency Room (ER) Visits
Description: The number of emergency room visits occurring during the treatment period will be compared between study groups.
Time Frame: Baseline through Week 26
Population: All participants that were randomized and received at least one dose of study medication and completed at least one follow-up.
Measure: Number; unit: Number of ER visits
Arm/Group | IDegLira | Basal-Bolus Insulin
Number analyzed (Participants) | 72 | 73
Number of ER visits | 14 | 12

26. Secondary Outcome: Number of Hospital Readmissions
Description: The number of hospital readmissions occurring during the treatment period will be compared between study groups.
Time Frame: Baseline through Week 26
Population: All participants who were randomized and received at least one dose of study medication and completed at least one follow-up.
Measure: Number; unit: Number of Hospital readmissions
Arm/Group | IDegLira | Basal-Bolus Insulin
Number analyzed (Participants) | 72 | 73
Number of Hospital readmissions | 0 | 4

27. Secondary Outcome: Total Daily Insulin Dose
Description: The total insulin dose measured in units per day will be compared between study groups.
Time Frame: Baseline, Week 26
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: units per day
Arm/Group | IDegLira | Basal-Bolus Insulin
Number analyzed (Participants) | 72 | 73
units per day
  Baseline | 24.56 (7.76) | 46.05 (20.79)
  26 weeks | 35.74 (17.53) | 75.65 (43.43)

ADVERSE EVENTS:
Time Frame: Duration of the study participation from enrollment up to 6 months
Arm/Group | IDegLira | Basal-Bolus Insulin
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/73
Serious Adverse Events (participants affected / at risk) | 14/72 | 12/73
Other Adverse Events (participants affected / at risk) | 30/72 | 13/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegLira (N=72) | Basal-Bolus Insulin (N=73)
Hospital Readmissions (General disorders) | 0 (0) | 4
Emergency Room Visits (General disorders) | 14 | 12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegLira (N=72) | Basal-Bolus Insulin (N=73)
Nausea (Gastrointestinal disorders) | 27 | 3 (3)
Vomiting (Gastrointestinal disorders) | 9 | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 13 (13) | 6
Diarrhea (Gastrointestinal disorders) | 8 (15) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/40/NCT03737240/Prot_SAP_000.pdf